CLINICAL TRIAL: NCT02741531
Title: The Effect of Partial Bladder Filling on Post-operative Time to Void in Minimally Invasive Gynecologic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121536
Record Dates: First submitted 2016-03-30; First posted 2016-04-18 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Hysterectomy; Myomectomy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients in this group will have their bladder filled with 150 cubic centimeters (cc) of saline solution prior to being moved to the PACU.
  Interventions: Other: Bladder filled with saline solution; Other: saline solution
- Control (No Intervention): patients in this group will have their bladders drained completely prior to being moved to the PACU as is the current standard of care.

INTERVENTIONS:
Other: Bladder filled with saline solution — Patients in this arm will have their bladders filled with 150 cc of saline solution.
  Arms: Intervention
Other: saline solution — Saline solution will be used to partially fill patients' bladders
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine if partially filling the bladder after laparoscopic/robotic gynecologic surgery (for benign disease) shortens the time required to spontaneously void for patients to determine if this subsequently shortens patient stay times in the Post Anesthesia Care Unit (PACU) following surgery. This intervention would be compared to the current standard of care, which involves removing the patient's Foley catheter with an empty bladder and then giving the patient up to 6 hours to void in the PACU.

DETAILED DESCRIPTION:
Patients undergoing laparoscopic/robotic hysterectomy or myomectomy who meet the study criteria will be contacted by the research assistant at a pre-operative visit. The risks and benefits of participation will be explained to them. If they choose to participate they will sign the consent form at that time.

At the time of the surgery, the research coordinator will open a sealed envelope containing the patient's assignment to partial bladder filling or no bladder filling. The research coordinator will then notify the surgeon via secure phone call or secure messaging service and the patient/subject will have their bladder partially filled or completely emptied as relayed to the surgeon at the end of the procedure in the Operating Room, unless there are issues of patient safety or operative complications. In the patients who are chosen for partial bladder filling, the bladder will be back-filled with 150 cc of normal saline and then the Foley catheter will be removed at the end of the procedure. In patients who have no bladder filling, the bladder will be completely emptied and then the Foley catheter will be removed. One of the providers who perform the gynecological surgical procedures will be responsible for back-filling or completely emptying the bladder with the Foley catheter.

The patients will be followed in the PACU to determine the time it takes for them to void. The will also be followed for any complications until they are four weeks post surgery. The electronic medical record will be examined to see if they have any complications reported at their post-operative visits or any readmissions to the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Hysterectomy or myomectomy planned for a benign gynecologic reason. (This means that there is no evidence of, or concern for, malignancy in the cervix, uterus, tubes or ovaries. Benign gynecologic reasons to have a hysterectomy include fibroids, abnormal uterine bleeding, endometriosis, and pelvic pain. Benign reason for myomectomy would be fibroids)
2. Patient is scheduled to have surgery with one of the minimally invasive gynecologic surgeons at George Washington University Hospital (GWUH)
3. Patient is planned for a robotic assisted total laparoscopic hysterectomy (RA-TLH) or a total laparoscopic hysterectomy (TLH) or robotic assisted or laparoscopic myomectomy.
4. Patient is capable of informed consent.
5. The patient has no baseline urinary disease.

Exclusion Criteria:

1. Hysterectomy or myomectomy is indicated for malignancy
2. Hysterectomy or myomectomy is not being performed via robotic or laparoscopic method
3. Patient is not capable of providing informed consent
4. Patient has urinary disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female or person with female sexual reproduction organs
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Time to Void | peri-operative
  the time (in minutes) between when the patient's foley is removed and when the patient is able to void in the PACU.

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Moawad G, Tyan P, Marfori C, Abi Khalil E, Park D. Effect of postoperative partial bladder filling after minimally invasive hysterectomy on postanesthesia care unit discharge and cost: a single-blinded, randomized controlled trial. Am J Obstet Gynecol. 2019 Apr;220(4):367.e1-367.e7. doi: 10.1016/j.ajog.2018.12.034. Epub 2019 Jan 9. PMID 30639089